CLINICAL TRIAL: NCT03466593
Title: Effekt av Prehabilitering Och Extra Tidig Mobilisering Efter öppen Pankreas Kirurgi
Brief Title: Effects of Prehabilitation and Early Mobilization for Patients Undergoing Pancreas Surgery.
Acronym: PreMob
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FoU i VGR: 238701
Record Dates: First submitted 2018-02-23; First posted 2018-03-15 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Pancreas Cancer
Keywords: Prehabilitation; Recovery; Complications
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: 1. A prospective cohort compared to historical controls
  2. A randomized, controlled, intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prospective cohort-prehabilitation (Experimental): A prehabilitation program including advice about diet, increased physical activity and cessation of smoking and drinking alcohol.
  Interventions: Other: Prehabilitation
- Retrospective cohort (Active Comparator): Routine care before the prehabilitation program was introduced
  Interventions: Other: Routine care
- Extra early mobilization (Experimental): Mobilization the day of surgery
  Interventions: Other: Extra early mobilization
- Traditional mobilization (Active Comparator): Routine care with mobilization the day after surgery
  Interventions: Other: Standard mobilization

INTERVENTIONS:
Other: Prehabilitation — Prehabilitation concerning eating, smoking, drinking and physical activity
  Arms: Prospective cohort-prehabilitation
Other: Routine care — Preoperative information
  Arms: Retrospective cohort
Other: Extra early mobilization — Mobilization the day of surgery
  Arms: Extra early mobilization
Other: Standard mobilization — Mobilization the day after surgery
  Arms: Traditional mobilization

SUMMARY:
Open upper gastrointestinal surgery includes surgery in the upper abdomen such as ventricular, duodenal, pancreatic and biliary tract surgery. After upper abdominal surgery there is a risk of gastrointestinal and cardiopulmonary complications. There is currently insufficient knowledge about the effect of prehabilitation and extra early postoperative mobilization in upper pancreatic surgery.

This study's aim is to evaluate the effect of prehabilitation and extra early mobilization.

The study includes two substudies:

1. A prospective cohort of 75 patients undergoing pancreatic surgery after a prehabilitation program will be compared to 75 historical controls. Primary outcome is postoperative complications.
2. A randomized controlled trial based on 72 patients undergoing pancreatic studying the effect of extra early rehabilitation. The intervention group will be mobilized to bedside, standing or sitting in armchair <6 hours after surgery, ie 3-4 hours after arrival at the Postoperative Department (PIVA). The control group will be mobilized according to routine i.e. the morning after surgery. Primary outcome is PaO2.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo pancreatic surgery

Exclusion Criteria in substudy b:

* Preoperative injury or disease making it impossible to perform the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | Whole study period from inclusion to one year after surgery
  Standardized complications according to register
PaO2 | The day before surgery to the first day after surgery
  Arterial oxygen pressure

SECONDARY OUTCOMES:
EORTC-module generic | Whole study period from inclusion to one year after surgery
  Quality of life, EORTC-QLQ-C30 (Range 30-124) Low values correspond to high quality of life
EORTC-module specific for pancreas cancer | Whole study period from inclusion to one year after surgery
  Quality of life QLQ-OG25 (Range 25- 100). Low values correspond to high quality of life
EORTC-module for fatigue | Whole study period from inclusion to one year after surgery
  Quality of Life FA-R13 (range 12- 48). Low values correspond to high quality of life
The Postoperative Recovery Profile | Whole study period from inclusion to one year after surgery
  Quality of recovery according to Allvin et al. 19 statements which are rated on a four grade scale fron no problem to major problem
Pancreatic cancer disease impact (PACADI) score | Whole study period from inclusion to one year after surgery
  Disease specific questionnaire, 8 statements rated on a visual analogue scale from 0 (no problem) to 10 (worst imaginable problem). Sum score are used for analysis (Range 0-80)
Spirometry | From inclusion (during preoperative information 1-14 days before surgery) to the first postoperative day after the operation
  Vital capacity
Lenght of stay | From the day before surgery to discharge from the hospital (app 7-14 days)
  Length of stay at the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Göteborg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fagevik Olsen M, Becovic S, Dean E. Short-term effects of mobilization on oxygenation in patients after open surgery for pancreatic cancer: a randomized controlled trial. BMC Surg. 2021 Apr 7;21(1):185. doi: 10.1186/s12893-021-01187-2. PMID 33827537